CLINICAL TRIAL: NCT02646579
Title: Effects of Dry Needling Using Spinal and Peripheral Sites Versus Peripheral Sites Only Among Individuals With Chronic Lower Extremity Conditions
Brief Title: Effects of Dry Needling Using Spinal and Peripheral Sites Versus Peripheral Sites Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marie Johanson, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00084277
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Plantar Fasciitis; Achilles Tendinitis; Patellofemoral Pain Syndrome
Keywords: Orthopedics
MeSH Terms: conditions — Fasciitis, Plantar; Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal and Peripheral Dry Needling (Experimental): Participants will receive dry needling to the low back and painful areas in the leg.
  Interventions: Procedure: Spinal and Peripheral Dry Needling
- Peripheral Dry Needling (Active Comparator): Participants will receive dry needling to painful areas in the leg.
  Interventions: Procedure: Peripheral Dry Needling

INTERVENTIONS:
Procedure: Spinal and Peripheral Dry Needling — Participants will be positioned lying flat and the relevant spinal level will be treated using a Seirin L- type 50 mm needle. The needle will be inserted to a depth no greater than three-quarters length of the needle for 30 seconds using a vertical pistoning technique and then statically up to 10 minutes.
  Arms: Spinal and Peripheral Dry Needling
Procedure: Peripheral Dry Needling — Participants will be positioned lying flat and the relevant peripheral points will be treated using a Seirin L- type 50 mm needle. The peripheral treatment site(s) will be determined by the physical therapist's palpation of active or latent trigger points or tender points. The needle will be inserted to a depth no greater than three-quarters length of the needle for 30 seconds using a vertical pistoning technique and then statically up to 10 minutes.
  Arms: Peripheral Dry Needling

SUMMARY:
The purpose of this study is to determine if dry needling both low back and extremity areas is more effective for reducing pain and improving strength, balance and functional performance among patients with chronic musculoskeletal conditions compared to dry needling of extremity areas only.

DETAILED DESCRIPTION:
This study will determine if spinal and peripheral dry needling sites results in decreased pain, increased muscle strength, increased proprioception and increased functional performance among individuals with chronic musculoskeletal conditions of the lower extremities, such as plantar fasciitis, Achilles tendinopathy, and patellofemoral pain syndrome. Specific aims are to determine if individuals with chronic musculoskeletal conditions of the lower extremities receiving dry needling to both spinal and peripheral sites exhibit differences in pain, muscle strength, proprioception, and unilateral hop test scores compared to individuals with chronic musculoskeletal conditions of the lower extremities receiving dry needling to peripheral sites only.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral chronic lower extremity musculoskeletal condition
* Ability to perform a unilateral one-quarter squat on involved side without pain
* Asymptomatic during walking

Exclusion Criteria:

* History of systemic neurological or arthritic condition
* History of bony or peripheral nerve trauma or surgery lower extremities
* No contraindications to dry needling
* Not currently receiving treatment for the chronic lower extremity musculoskeletal condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Level assessed using the Visual Analogue Scale (VAS) | Baseline, Visit 2 (Up to 7 days)
  Pain level will be assessed using the Visual Analogue Scale (VAS). The pain VAS is a self-reported, single-item scale that ranks pain level from no pain to worst imaginable pain on a single scale line. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the participant's mark, providing a range of scores from 0-100.

SECONDARY OUTCOMES:
Change in Muscle Strength of Hip Abductors assessed using a dynamometer | Baseline, Visit 2 (Up to 7 days)
  The strength of the hip abductors will be assessed using a dynamometer. The subjects will be asked to exert maximal force against the dynamometer and the reading is recorded. Scores are based on force production in kilograms or pounds; kilograms (0-90), pounds (0-200). Higher pressure scores indicate better muscle strength of the hip abductor muscles.
Change in Muscle Strength of Knee Extensors/Flexors assessed using a dynamometer | Baseline, Visit 2 (Up to 7 days)
  The strength of the knee extensors/flexors will be assessed using a dynamometer. The subjects will be asked to exert maximal force against the dynamometer and the reading is recorded. Scores are based on force production in kilograms or pounds; kilograms (0-90), pounds (0-200). Higher pressure scores indicate better muscle strength of the knee extensor/flexor muscles.
Change in Muscle Strength of Ankle Dorsiflexors/Platarflexors assessed using a dynamometer | Baseline, Visit 2 (Up to 7 days)
  The strength of the ankle dorsiflexors/platarflexors will be assessed using a dynamometer. The subjects will be asked to exert maximal force against the dynamometer and the reading is recorded. Scores are based on force production in kilograms or pounds; kilograms (0-90), pounds (0-200). Higher pressure scores indicate better muscle strength of the ankle dorsiflexor/platarflexor muscles.
Change in Unilateral Hop Distance | Baseline, Visit 2 (Up to 7 days)
  Participants will perform a single leg hop for distance with each lower extremity. After demonstration, each participant will be allowed 1 trial per leg. Beginning with the toes immediately behind the starting line, participants will perform one hop to complete a trial. The hop will be measured from the starting line to the end of the toes after completion of a trial. Each limb will be tested two times with the maximal distance scored for each limb. Scores will be recorded as absolute distance (in centimeters). An increase in the score (distance covered) from baseline visit to visit 2 indicates better functional performance of the muscles.
Change in Single-limb Standing Balance Test Time | Baseline, Visit 2 (Up to 7 days)
  Participants will attempt to balance themselves within a defined area on a single limb. The maximum amount of time will be calculated both with and without their eyes closed. The opposite leg must be out in front of the participant fully extended and will not be allowed to touch any part of the body. The test will be timed, up to two minutes, on each limb with two trials on either side.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Johanson, PhD, Principal Investigator — Emory University
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States